CLINICAL TRIAL: NCT05769153
Title: A Phase 1/2 Two-Stage Dose Escalation and Randomized Parallel-Group Study to Evaluate the Safety, Preliminary Treatment Effects, and Durability of AR-14034 Sustained Release Implant Compared to Intravitreal Anti-Vascular Endothelial Growth Factor Treatment in Participants With Neovascular Age-Related Macular Degeneration
Brief Title: Study of AR-14034 in Participants With Neovascular Age-Related Macular Degeneration (nAMD)
Acronym: NOVA-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RTE888-E001
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Neovascular Age-related Macular Degeneration (nAMD)
Keywords: nAMD; retina; eyes; ophthalmology
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: Stage 1 will enroll 2 cohorts. Stage 2 will enroll 3 treatment arms.
Who Masked: Participant, Investigator
Masking Description: Stage 1 is open label. Stage 2 is double-masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1 (Stage 1) (Experimental): One intravitreal (IVT) injection of aflibercept 2 mg at Week -1 and one IVT insertion of AR-14034 SR lower dose at Baseline. Up to one retreatment with AR-14034 SR will be administered between Weeks 4 and 36 according to protocol-specified disease activity criteria.
  Interventions: Drug: AR-14034 SR implant lower dose; Drug: Aflibercept Injection
- Cohort 2 (Stage 1) (Experimental): One IVT injection of aflibercept 2 mg at Week -1 and one IVT insertion of AR-14034 SR higher dose at Baseline. Up to one retreatment with AR-14034 SR will be administered between Weeks 4 and 36 according to protocol-specified disease activity criteria.
  Interventions: Drug: AR-14034 SR implant higher dose; Drug: Aflibercept Injection
- AR-14034 SR one injection (Stage 2) (Experimental): One IVT injection of aflibercept 2 mg at Baseline, Week 4, and Week 8, with one IVT insertion of AR-14034 SR at Week 2. Sham procedures will be performed between Baseline and Week 52 when other arms are receiving scheduled treatment injections.
  Interventions: Drug: AR-14034 SR implant; Drug: Aflibercept Injection; Drug: Sham procedure
- AR-14034 SR two injections (Stage 2) (Experimental): One IVT injection of aflibercept 2 mg at Baseline, Week 4, and Week 8, with IVT insertions of AR-14034 SR at Week 2 and Week 6. Sham procedures will be performed between Baseline and Week 52 when other arms are receiving scheduled treatment injections.
  Interventions: Drug: AR-14034 SR implant; Drug: Aflibercept Injection; Drug: Sham procedure
- Aflibercept (Stage 2) (Active Comparator): One IVT injection of aflibercept 2 mg at Baseline, Week 4, Week 8, Week 16, Week 24, Week 32, Week 40, and Week 48. Sham procedures will be performed between Baseline and Week 52 when other arms are receiving scheduled treatment injections.
  Interventions: Drug: Aflibercept Injection; Drug: Sham procedure

INTERVENTIONS:
Drug: AR-14034 SR implant lower dose — AR-14034 SR administered as an intravitreal implant
  Arms: Cohort 1 (Stage 1)
Drug: AR-14034 SR implant higher dose — AR-14034 SR administered as an intravitreal implant
  Arms: Cohort 2 (Stage 1)
Drug: AR-14034 SR implant — AR-14034 SR administered as an intravitreal implant
  Arms: AR-14034 SR one injection (Stage 2); AR-14034 SR two injections (Stage 2)
Drug: Aflibercept Injection — Aflibercept administered as a 2 milligram (mg) intravitreal injection
Drug: Sham procedure — Needleless syringe used to simulate an intravitreal injection
  Arms: AR-14034 SR one injection (Stage 2); AR-14034 SR two injections (Stage 2); Aflibercept (Stage 2)

SUMMARY:
The primary purpose of this study is to evaluate the safety and durability of single- and repeat administration of AR-14034 Sustained Release (SR) in subjects with neovascular age-related macular degeneration (nAMD).

DETAILED DESCRIPTION:
This study will be conducted in two stages. Stage 1 is a 48-week, dose-escalation, open-label evaluation of AR-14034 SR. Two cohorts will be enrolled, for an approximate total of 10 subjects. Subjects will receive AR-14034 SR in one of two dose levels and attend visits through Week 48 for assessment of safety and preliminary treatment effects.

Stage 2 is a 56-week (plus extension) double-masked, active comparator, randomized, parallel group evaluation of AR-14034 SR compared with aflibercept. Approximately 130 subjects will be enrolled and randomized 2:2:1 to AR-14034 SR one injection, AR-14034 SR two injections, or aflibercept dosed as labelled. Subjects will attend visits through Week 56 for assessment of safety and treatment effects. A 16-week open label extension phase will be conducted thereafter.

ELIGIBILITY:
Key Inclusion Criteria [Stage 1 and Stage 2]:

* Presence of an active choroidal neovascularization (CNV) lesion secondary to age-related macular degeneration (AMD);
* Best corrected visual acuity (BCVA) between 80 and 35 letters (20/25 to 20/200 Snellen equivalent) in the study eye;
* BCVA greater than 20 letters (approximately 20/400 Snellen equivalent) in the non-study eye;
* Media clarity and pupillary dilation in the study eye sufficient for all planned study procedures;
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol;
* Other protocol-specified inclusion criteria may apply.

[Stage 1]:

* Greater than or equal to 3 and less than or equal to 6 prior treatments of an ocular anti-VEGF medication within the 8 months prior to Screening in the study eye, with demonstrated anatomic response, as assessed by the Investigator.

[Stage 2]:

* Treatment-naïve, or diagnosis of exudative neovascular age-related macular degeneration (nAMD) in the study eye.

Key Exclusion Criteria [Stage 1 and Stage 2]:

* History or current ocular disease in the study eye other than nAMD, that, might require medical or surgical intervention during the study;
* Structural damage to the macula that is likely to preclude improvement in visual acuity in the study eye after resolution of the nAMD;
* Any active intraocular or periocular infection or active intraocular inflammation;
* Treatment with ocular anti-VEGF product in the study eye within 28 days before Week 1 [Stage 1] or within 56 days before Screening [Stage 2].
* Uncontrolled glaucoma in the study eye;
* Uncontrolled blood pressure;
* Females of child-bearing potential who are pregnant, intending to become pregnant, nursing, or who are not willing to use an acceptable form of contraception for the duration of the study;
* Other protocol-specified exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in ETDRS BCVA at the average across two visits, Weeks 44 and 48 (Stage 2) | Baseline, Week 44, Week 48
  Visual acuity will be measured after manifest refraction using Early Treatment of Diabetic Retinopathy Study (ETDRS) letter charts in a 4-meter lane under standard illumination. Best corrected visual acuity (BCVA) will be recorded as the number of letters read correctly. The difference between the average across Weeks 44 and 48, and the baseline visit will be reported. One eye (study eye) will contribute to the analysis.

SECONDARY OUTCOMES:
Mean change from baseline in ETDRS BCVA by visit (Stage 2) | Baseline to Week 56
  Visual acuity will be measured after manifest refraction using ETDRS letter charts in a 4-meter lane under standard illumination. BCVA will be recorded as the number of letters read correctly. The difference between a given post-baseline visit and the baseline visit will be reported. One eye (study eye) will contribute to the analysis.
Mean change from baseline in Central Subfield Thickness (CST) by visit (Stage 2) | Baseline to Week 56
  Central subfield thickness (CST) will be assessed using spectral domain optical coherence tomography (SD-OCT) imaging and measured in micrometers. The difference between a given post-baseline visit and the baseline visit will be reported. One eye (study eye) will contribute to the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Director of Clinical Development, Alcon, Study Director — Alcon Research, LLC
Locations (42):
- United States (42):
  - Trinity Research Group, Dothan, Alabama
  - Associated Retina Consultants - Gilbert, Gilbert, Arizona
  - Associated Retina Consultants - Phoenix, Phoenix, Arizona
  - Retina Associates of SW PC, Tucson, Arizona
  - The Retina Partners, Encino, California
  - Retina Associates of Orange County, Laguna Hills, California
  - Northern California Retina Vitreous Associates Medical Group, Mountain View, California
  - Eye Research Foundation, Newport Beach, California
  - Azul Vision Pasadena, Pasadena, California
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - Retina Group of New England | Waterford, Waterford, Connecticut
  - Florida Retina Institute, Jacksonville, Florida
  - Mid Florida Eye Center, Mt. Dora, Florida
  - Florida Retina Institute, Orlando, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Eye Associates of Pinellas, Pinellas Park, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - Thomas Eye Group Main Office, Sandy Springs, Georgia
  - University Retina and Macula Associates, PC, Oak Forest, Illinois
  - Twin Cities Eye Consultants, Coon Rapids, Minnesota
  - Mississippi Retina Associates, Madison, Mississippi
  - Vision Research Center Eye Associates of New Mexico, Albuquerque, New Mexico
  - NYC Retina - Queens, Forest Hills, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Verum Research, LLC, Eugene, Oregon
  - Erie Retina Research, Erie, Pennsylvania
  - MidAtlantic Retina Research, Philadelphia, Pennsylvania
  - Retina Consultants of Carolina, Greenville, South Carolina
  - Carolina Eyecare Physicians LLC, Mt. Pleasant, South Carolina
  - Retina Research Institute of Texas, Abilene, Texas
  - Texas Retina Associates - Arlington, Arlington, Texas
  - Austin Research Center for Retina, Austin, Texas
  - Austin Retina Associates, Austin, Texas
  - Austin Clinical Research, LLC, Austin, Texas
  - Star Vision Research, Burleson, Texas
  - Texas Retina Associates, Dallas, Texas
  - Berkeley Eye Center, Houston, Texas
  - Retina Consultants of Texas - San Antonio, San Antonio, Texas
  - Austin Retina Associates (San Marcos), San Marcos, Texas
  - Retina Research Center of Southern Utah, St. George, Utah
  - Pacific Northwest Retina, Burlington, Washington

IPD SHARING:
Plan to Share IPD: No